CLINICAL TRIAL: NCT02238054
Title: French Observatory Evaluating the Use of Intracoronary Prosthesis ABSORB BVS
Acronym: FRANCE-ABSORB
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 14249
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Intracoronary Angioplasty
Keywords: Cardiology; Intracoronary angioplasty; Bioresorbable stent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ABSORB BVS: All patients with a coronary angioplasty procedure and the implantation of at least one ABSORB BVS

SUMMARY:
Observational Study, French, prospective, multicenter rated using intravascular prosthesis ABSORB BVS.

ABSORB BVS is a prosthesis of a new type. This study will prospectively evaluate all procedures for coronary angioplasty with implantation of at least one BVS with a clinical follow-up of all patients implanted with ABSORB BVS. This national observatory will collect all the events related to product and / or to procedure

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated to the National Health Insurance Scheme
* Patient able to assess and understand the risks, benefits and alternative treatments laying of ABSORB, to agree to participate in the study (by signing the informed consent after having read the newsletter)
* Patients for whom a procedure is performed coronary angioplasty with implantation of at least one BVS.
* Patient allowing the follow-up as defined in the study

Exclusion Criteria:

* Pregnant patient
* Patient that can not give informed consent
* Patient with in-stent restenosis or saphenous vein bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the departments of Cardiology, from French health institutions, who are authorized to implement, may participate in the observatory.
  It is estimated that this procedure will be performed by 50 to 60 sites performing the installation of BVS. The list of centers is scalable, their number can be expected to increase.
Sampling Method: Non-Probability Sample
Enrollment: 2072 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events at 1 year | 1 year
  At 1 year of follow-up, to evaluate the rate of MACE (Major Adverse Cardiac Events) defined as follows:
  * Death from cardiac causes
  * Myocardial Infarction
  * Rates of target lesion revascularization (TLR) of ischemic origin (ID-TLR)
  * Surgery unscheduled bypass graft (CABG)

SECONDARY OUTCOMES:
Target vessel revascularization at 1 year | 1 year
  At 1 year of follow-up, to evaluate the rate of target vessel revascularization (TVR)
Rate of stent thrombosis at 1 year | 1 year
  At 1 year of follow-up, to evaluate the rate of stent thrombosis as ARC definitions :
  * acute, subacute, late
  * probable or undoubted

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Saint Hilaire, Rouen, France

REFERENCES:
- [Background] Sigwart U, Puel J, Mirkovitch V, Joffre F, Kappenberger L. Intravascular stents to prevent occlusion and restenosis after transluminal angioplasty. N Engl J Med. 1987 Mar 19;316(12):701-6. doi: 10.1056/NEJM198703193161201. PMID 2950322
- [Background] Gruntzig AR, Senning A, Siegenthaler WE. Nonoperative dilatation of coronary-artery stenosis: percutaneous transluminal coronary angioplasty. N Engl J Med. 1979 Jul 12;301(2):61-8. doi: 10.1056/NEJM197907123010201. PMID 449946
- [Background] Serruys PW, de Jaegere P, Kiemeneij F, Macaya C, Rutsch W, Heyndrickx G, Emanuelsson H, Marco J, Legrand V, Materne P, et al. A comparison of balloon-expandable-stent implantation with balloon angioplasty in patients with coronary artery disease. Benestent Study Group. N Engl J Med. 1994 Aug 25;331(8):489-95. doi: 10.1056/NEJM199408253310801. PMID 8041413
- [Background] Serruys PW, Kutryk MJ, Ong AT. Coronary-artery stents. N Engl J Med. 2006 Feb 2;354(5):483-95. doi: 10.1056/NEJMra051091. No abstract available. PMID 16452560
- [Background] Morice MC, Serruys PW, Sousa JE, Fajadet J, Ban Hayashi E, Perin M, Colombo A, Schuler G, Barragan P, Guagliumi G, Molnar F, Falotico R; RAVEL Study Group. Randomized Study with the Sirolimus-Coated Bx Velocity Balloon-Expandable Stent in the Treatment of Patients with de Novo Native Coronary Artery Lesions. A randomized comparison of a sirolimus-eluting stent with a standard stent for coronary revascularization. N Engl J Med. 2002 Jun 6;346(23):1773-80. doi: 10.1056/NEJMoa012843. PMID 12050336
- [Background] Abbott JD, Voss MR, Nakamura M, Cohen HA, Selzer F, Kip KE, Vlachos HA, Wilensky RL, Williams DO. Unrestricted use of drug-eluting stents compared with bare-metal stents in routine clinical practice: findings from the National Heart, Lung, and Blood Institute Dynamic Registry. J Am Coll Cardiol. 2007 Nov 20;50(21):2029-36. doi: 10.1016/j.jacc.2007.07.071. PMID 18021868
- [Background] Ormiston JA, Serruys PW, Regar E, Dudek D, Thuesen L, Webster MW, Onuma Y, Garcia-Garcia HM, McGreevy R, Veldhof S. A bioabsorbable everolimus-eluting coronary stent system for patients with single de-novo coronary artery lesions (ABSORB): a prospective open-label trial. Lancet. 2008 Mar 15;371(9616):899-907. doi: 10.1016/S0140-6736(08)60415-8. PMID 18342684
- [Background] Serruys PW, Ormiston JA, Onuma Y, Regar E, Gonzalo N, Garcia-Garcia HM, Nieman K, Bruining N, Dorange C, Miquel-Hebert K, Veldhof S, Webster M, Thuesen L, Dudek D. A bioabsorbable everolimus-eluting coronary stent system (ABSORB): 2-year outcomes and results from multiple imaging methods. Lancet. 2009 Mar 14;373(9667):897-910. doi: 10.1016/S0140-6736(09)60325-1. PMID 19286089
- [Background] Serruys PW, Onuma Y, Ormiston JA, de Bruyne B, Regar E, Dudek D, Thuesen L, Smits PC, Chevalier B, McClean D, Koolen J, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Miquel-Hebert K, Rapoza R, Garcia-Garcia HM. Evaluation of the second generation of a bioresorbable everolimus drug-eluting vascular scaffold for treatment of de novo coronary artery stenosis: six-month clinical and imaging outcomes. Circulation. 2010 Nov 30;122(22):2301-12. doi: 10.1161/CIRCULATIONAHA.110.970772. Epub 2010 Nov 15. PMID 21098436
- [Background] Serruys PW, Onuma Y, Dudek D, Smits PC, Koolen J, Chevalier B, de Bruyne B, Thuesen L, McClean D, van Geuns RJ, Windecker S, Whitbourn R, Meredith I, Dorange C, Veldhof S, Hebert KM, Sudhir K, Garcia-Garcia HM, Ormiston JA. Evaluation of the second generation of a bioresorbable everolimus-eluting vascular scaffold for the treatment of de novo coronary artery stenosis: 12-month clinical and imaging outcomes. J Am Coll Cardiol. 2011 Oct 4;58(15):1578-88. doi: 10.1016/j.jacc.2011.05.050. PMID 21958884
- [Background] Dudek D, Onuma Y, Ormiston JA, Thuesen L, Miquel-Hebert K, Serruys PW. Four-year clinical follow-up of the ABSORB everolimus-eluting bioresorbable vascular scaffold in patients with de novo coronary artery disease: the ABSORB trial. EuroIntervention. 2012 Jan;7(9):1060-1. doi: 10.4244/EIJV7I9A168. PMID 21959320
- [Background] Ormiston J, Webster M. Absorbable coronary stents. Lancet. 2007 Jun 2;369(9576):1839-1840. doi: 10.1016/S0140-6736(07)60829-0. No abstract available. PMID 17544749
- [Background] Ramcharitar S, Serruys PW. Fully biodegradable coronary stents : progress to date. Am J Cardiovasc Drugs. 2008;8(5):305-14. doi: 10.2165/00129784-200808050-00003. PMID 18828642
- [Background] Macaya C, Moreno R. Bioabsorbable drug-eluting stents: the future of coronary angioplasty? Nat Clin Pract Cardiovasc Med. 2008 Oct;5(10):598-9. doi: 10.1038/ncpcardio1306. Epub 2008 Aug 5. PMID 18679382
- [Background] Colombo A, Sharp AS. The bioabsorbable stent as a virtual prosthesis. Lancet. 2009 Mar 14;373(9667):869-70. doi: 10.1016/S0140-6736(09)60521-3. No abstract available. PMID 19286066
- [Background] Ormiston JA, Serruys PW. Bioabsorbable coronary stents. Circ Cardiovasc Interv. 2009 Jun;2(3):255-60. doi: 10.1161/CIRCINTERVENTIONS.109.859173. No abstract available. PMID 20031723
- [Background] Onuma Y, Piazza N, Ormiston JA, Serruys PW. Everolimus-eluting bioabsorbable stent--Abbot Vascular programme. EuroIntervention. 2009 Dec 15;5 Suppl F:F98-F102. doi: 10.4244/EIJV5IFA17. No abstract available. PMID 22100687
- [Background] Oberhauser JP, Hossainy S, Rapoza RJ. Design principles and performance of bioresorbable polymeric vascular scaffolds. EuroIntervention. 2009 Dec 15;5 Suppl F:F15-22. doi: 10.4244/EIJV5IFA3. PMID 22100671
- [Background] Onuma Y, Serruys PW, Ormiston JA, Regar E, Webster M, Thuesen L, Dudek D, Veldhof S, Rapoza R. Three-year results of clinical follow-up after a bioresorbable everolimus-eluting scaffold in patients with de novo coronary artery disease: the ABSORB trial. EuroIntervention. 2010 Sep;6(4):447-53. doi: 10.4244/EIJ30V6I4A76. PMID 20884431
- [Background] Bittl JA. Bioresorbable stents: the next revolution. Circulation. 2010 Nov 30;122(22):2236-8. doi: 10.1161/CIRCULATIONAHA.110.988469. Epub 2010 Nov 15. No abstract available. PMID 21098438
- [Background] Diletti R, Onuma Y, Farooq V, Gomez-Lara J, Brugaletta S, van Geuns RJ, Regar E, de Bruyne B, Dudek D, Thuesen L, Chevalier B, McClean D, Windecker S, Whitbourn R, Smits P, Koolen J, Meredith I, Li D, Veldhof S, Rapoza R, Garcia-Garcia HM, Ormiston JA, Serruys PW. 6-month clinical outcomes following implantation of the bioresorbable everolimus-eluting vascular scaffold in vessels smaller or larger than 2.5 mm. J Am Coll Cardiol. 2011 Jul 12;58(3):258-64. doi: 10.1016/j.jacc.2011.02.052. PMID 21737016
- [Background] Gori T, Schulz E, Hink U, Wenzel P, Post F, Jabs A, Munzel T. Early outcome after implantation of Absorb bioresorbable drug-eluting scaffolds in patients with acute coronary syndromes. EuroIntervention. 2014 Jan 22;9(9):1036-41. doi: 10.4244/EIJV9I9A176. PMID 23999237
- [Background] Simsek C, Magro M, Onuma Y, Boersma E, Smits P, Dorange C, Veldhof S, Regar E, Serruys PW, van Geuns RJ. Procedural and clinical outcomes of the Absorb everolimus-eluting bioresorbable vascular scaffold: one-month results of the Bioresorbable vascular Scaffold Evaluated At Rotterdam Cardiology Hospitals (B-SEARCH). EuroIntervention. 2014 Jun;10(2):236-40. doi: 10.4244/EIJV10I2A38. PMID 23999210
- [Background] Meincke F, Kuck KH, Bergmann MW. Delivery of a bioresorbable vascular scaffold to complex lesions. Catheter Cardiovasc Interv. 2014 Nov 1;84(5):774-8. doi: 10.1002/ccd.25105. Epub 2014 Jul 30. PMID 23907893
- [Background] Kajiya T, Liang M, Sharma RK, Lee CH, Chan MY, Tay E, Chan KH, Tan HC, Low AF. Everolimus-eluting bioresorbable vascular scaffold (BVS) implantation in patients with ST-segment elevation myocardial infarction (STEMI). EuroIntervention. 2013 Aug 22;9(4):501-4. doi: 10.4244/EIJV9I4A80. PMID 23687101
- [Background] Gogas BD, Bourantas CV, Garcia-Garcia HM, Onuma Y, Muramatsu T, Farooq V, Diletti R, van Geuns RJ, De Bruyne B, Chevalier B, Thuesen L, Smits PC, Dudek D, Koolen J, Windecker S, Whitbourn R, McClean D, Dorange C, Miquel-Hebert K, Veldhof S, Rapoza R, Ormiston JA, Serruys PW. The edge vascular response following implantation of the Absorb everolimus-eluting bioresorbable vascular scaffold and the XIENCE V metallic everolimus-eluting stent. First serial follow-up assessment at six months and two years: insights from the first-in-man ABSORB Cohort B and SPIRIT II trials. EuroIntervention. 2013 Oct;9(6):709-20. doi: 10.4244/EIJV9I6A115. PMID 23628499
- [Background] Diletti R, Serruys PW, Farooq V, Sudhir K, Dorange C, Miquel-Hebert K, Veldhof S, Rapoza R, Onuma Y, Garcia-Garcia HM, Chevalier B. ABSORB II randomized controlled trial: a clinical evaluation to compare the safety, efficacy, and performance of the Absorb everolimus-eluting bioresorbable vascular scaffold system against the XIENCE everolimus-eluting coronary stent system in the treatment of subjects with ischemic heart disease caused by de novo native coronary artery lesions: rationale and study design. Am Heart J. 2012 Nov;164(5):654-63. doi: 10.1016/j.ahj.2012.08.010. PMID 23137495
- [Background] Diletti R, Farooq V, Girasis C, Bourantas C, Onuma Y, Heo JH, Gogas BD, van Geuns RJ, Regar E, de Bruyne B, Dudek D, Thuesen L, Chevalier B, McClean D, Windecker S, Whitbourn RJ, Smits P, Koolen J, Meredith I, Li X, Miquel-Hebert K, Veldhof S, Garcia-Garcia HM, Ormiston JA, Serruys PW. Clinical and intravascular imaging outcomes at 1 and 2 years after implantation of absorb everolimus eluting bioresorbable vascular scaffolds in small vessels. Late lumen enlargement: does bioresorption matter with small vessel size? Insight from the ABSORB cohort B trial. Heart. 2013 Jan;99(2):98-105. doi: 10.1136/heartjnl-2012-302598. Epub 2012 Oct 31. PMID 23118346
- [Background] Garcia-Garcia HM, Schultz C, Duckers E, Regar E, Ligthart J, Serruys PW, van Geuns RJ. Five-year follow-up of the ABSORB bioresorbable everolimus-eluting vascular scaffold system: multimodality imaging assessment. EuroIntervention. 2013 Feb 22;8(10):1126-7. doi: 10.4244/EIJV8I10A187. No abstract available. PMID 23014900
- [Background] Gogas BD, Farooq V, Onuma Y, Serruys PW. The ABSORB bioresorbable vascular scaffold: an evolution or revolution in interventional cardiology? Hellenic J Cardiol. 2012 Jul-Aug;53(4):301-9. No abstract available. PMID 22796817
- [Background] Brugaletta S, Garcia-Garcia HM, Onuma Y, Serruys PW. Everolimus-eluting ABSORB bioresorbable vascular scaffold: present and future perspectives. Expert Rev Med Devices. 2012 Jul;9(4):327-38. doi: 10.1586/erd.12.17. Epub 2012 Mar 16. PMID 22420293
- [Background] Gomez-Lara J, Diletti R, Brugaletta S, Onuma Y, Farooq V, Thuesen L, McClean D, Koolen J, Ormiston JA, Windecker S, Whitbourn R, Dudek D, Dorange C, Veldhof S, Rapoza R, Regar E, Garcia-Garcia HM, Serruys PW. Angiographic maximal luminal diameter and appropriate deployment of the everolimus-eluting bioresorbable vascular scaffold as assessed by optical coherence tomography: an ABSORB cohort B trial sub-study. EuroIntervention. 2012 Jun 20;8(2):214-24. doi: 10.4244/EIJV8I2A35. PMID 22030265
- [Background] Sarno G, Bruining N, Onuma Y, Garg S, Brugaletta S, De Winter S, Regar E, Thuesen L, Dudek D, Veldhof S, Dorange C, Garcia-Garcia HM, Ormiston JA, Serruys PW. Morphological and functional evaluation of the bioresorption of the bioresorbable everolimus-eluting vascular scaffold using IVUS, echogenicity and vasomotion testing at two year follow-up: a patient level insight into the ABSORB A clinical trial. Int J Cardiovasc Imaging. 2012 Jan;28(1):51-8. doi: 10.1007/s10554-010-9769-y. Epub 2011 Jan 7. PMID 21213050
- [Result] Cayla G, Koning R, Fajadet J, Sainsous J, Carrie D, Elhadad S, Tarragano F, Lefevre T, Ranc S, Ghostine S, Garot P, Marco F, Maillard L, Motreff P, Le Breton H; FRANCE ABSORB investigators. Percutaneous coronary interventions with the Absorb Bioresorbable vascular scaffold in real life: 1-year results from the FRANCE ABSORB registry. Arch Cardiovasc Dis. 2019 Feb;112(2):113-123. doi: 10.1016/j.acvd.2018.09.007. Epub 2019 Jan 7. PMID 30630761
- [Result] Lhermusier T, Carrie D, Cayla G, Fajadet J, Sainsous J, Elhadad S, Tarragano F, Chevalier B, Ranc S, Curinier C, Le Breton H, Koning R; FRANCE ABSORB Investigators. Three-year clinical outcomes with the ABSORB bioresorbable vascular scaffold in real life: Insights from the France ABSORB registry. Catheter Cardiovasc Interv. 2021 Sep;98(3):511-519. doi: 10.1002/ccd.29369. Epub 2020 Nov 19. PMID 33211387